CLINICAL TRIAL: NCT03992222
Title: Prevention of the Older Adult's Loss of Autonomy at Home Through a Physical Exercise Program Targeted at Adapted Muscle Strengthening Devices
Brief Title: Prevention of the Older Adult's Loss of Autonomy at Home Through a Targeted Physical Exercise Program
Acronym: PREPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K 170 919
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-01

CONDITIONS: Autonomy of Older People

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- administration of a physical exercise programme (Experimental): administration of a Physical exercise program for 24 weeks.
  Interventions: Device: Physical exercise programs PEP targeted on appropriate muscle strengthening devices allows
- control (No Intervention)

INTERVENTIONS:
Device: Physical exercise programs PEP targeted on appropriate muscle strengthening devices allows — administration of a Physical exercise program for 24 weeks.The participants will be followed at the 24 and 52nd weeks.
  Arms: administration of a physical exercise programme

SUMMARY:
Physical exercise program (PEP) have demonstrated their benefit to the health of older people. They are effective in functional performance and in the incidence and severity of falls.

We hypothesize that intervention with targeted Physical exercise programs PEP on appropriate muscle strengthening devices allows, through its action on the muscle, to slow down the loss of autonomy in the elderly living in the home. Our main objective is to evaluate the impact of a PEP, targeted on adapted muscle strengthening devices, on the loss of autonomy for the acts of daily life in the person aged over 70 living at home.

DETAILED DESCRIPTION:
The elderly will be identified during their call in the home centers of the town halls to get a housekeeper. After information, inclusion and randomization into two groups in the consultation site, the intervention group volunteers will follow the PEP for 24 weeks; the control group volunteers will receive a counseling booklet. Both groups will be followed at week 24 and 52.

ELIGIBILITY:
Inclusion Criteria:

* People over 70 years old
* Living at home
* With at least one instrumental activity of altered daily life (a disturbed criterion on the IADL scale) and making a request to set up a housekeeper.
* Major, able to give their consent
* Having signed the informed consent
* Affiliation to a social security scheme,

Exclusion Criteria:

* Surgical procedure within 6 months on the hip or knee,
* myocardial infarction or cerebrovascular accident diagnosed within 6 months,
* Respiratory insufficiency requiring long-term oxygen therapy
* Heart failure requiring hospitalization in the previous month or considered severe by the cardiologist
* Known or disabling muscle or joint pathology
* Subject benefiting from rehabilitation through physiotherapy sessions in progress or not wishing to stop physical exercise workshops
* Subject already in loss of autonomy for the ADL
* Life expectancy of less than 6 months any cause combined

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of people without activities of daily living (LDA) assessed by the 12-month Katz questionnaire in the intervention group compared to the control group. | 12 months
  To evaluate the impact of targeted PEEP on appropriate muscle strengthening devices, on the loss of autonomy for the acts of daily life in the person over 70 years old living at home

CONTACTS AND LOCATIONS:
Overall Officials: Véronique FRANCOIS, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital René Muret, Sevran, France